CLINICAL TRIAL: NCT00791531
Title: Phase 1 Assessment of Safety and Pharmacokinetics of a Low Dose of Methotrexate in Healthy Adult Male Kenyan Volunteers
Brief Title: Assessment of Safety and Pharmacokinetics of a Low Dose of Methotrexate in Healthy Adult Male Kenyan Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSC1464
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Malaria
Keywords: Methotrexate; Malaria
MeSH Terms: conditions — Malaria | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate (Experimental): Oral methotrexate 5mg once daily for 5 consecutive days
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Oral methotrexate 5mg once daily for 5 consecutive days
  Other Names: Methotrexate Lerdele

SUMMARY:
Previous investigations indicate that methotrexate, an old anticancer drug, could be used at low doses to treat malaria. This is a phase I evaluation to assess the safety and pharmacokinetic profile of this drug in healthy adult male Kenyan volunteers.

DETAILED DESCRIPTION:
Background Currently the control of malaria rests on the use of chemotherapy. However, the development of resistance to common used drugs represents a major public concern. Thus, the investigators need to develop new and cheap drugs. The investigators have discovered that the old drug methotrexate (MTX), which is used in the treatment of cancer and rheumatoid arthritis (RA), is very active against malaria parasites, including those that are resistant to existing antimalarials.

In the treatment of RA, MTX is used weekly at a low dose for several years. At dose, MTX is safe and well tolerated in human and children. This low dose of MTX will also kill malaria parasite in human. Thus, want to study MTX as an antimalarial. As part of this study, the investigators need to establish whether at the dose the investigators want it, 5 mg per days for 5 days, the drug is safe and well tolerated in 25 Kenyan adult volunteers. This result of this study will inform us on the use of MTX in the treatment of malaria in children.

What questions are the investigators trying to answer?

The investigators are trying to assess the safety of 5mg dose per day for 5

Where is the study taking place, how many people does it involve and how are they selected?

The study is taking place at KEMRI, Centre for Clinical Research, Nairobi. The study will involve 25 healthy adults.

What does the study involve for those who are taking part? Healthy adult males will be invited to join the study. A small blood sample will be collected from the arm to assess how the body is responding, the state of blood, liver and kidney functioning before and after the administration of the drug. This sample will also be used to rule out the presence of other infections such as HIV and Hepatitis.

Study patients will be given MTX every day for 5 days. During the days of Hospitalization patients will be assessed by physical examination, and tests to check for their liver function on day 1 and 5. Patients will then be followed up for a minimum of 42 days and will be seen at the clinics on days 7, 14, 28 and 42. The state of blood, liver and kidney will be done only before starting treatment and on day 28. Patients will also be required to undergo more samples to assess the level of the drug in their blood at different times from starting of treatment.

What are the benefits and risks/costs of the study for those involved Study subjects will receive full medical consultation and treatment through-out the study period. Long term benefits could be the addition of MTX to the list of antimalaria drugs available for treatment of non serious malaria. During the follow up period they will have the opportunity for their health to be followed up closely with a dedicated team of clinicians.

MTX has been used extensively at low dose in the treatment of RA. The drug is safe and well tolerated in human and children. However, when used on a chronic basis, few adverse reactions have so far been reported, mostly gastrointestinal upsets associated with nausea and vomiting. The risk this sign to occur is very small since we will use the drug for 5 days only.

How will the study benefit society? This study may help in development of MTX as a cheap, safe and easy to use drug in the treatment of malaria to add to the already available list of drugs.

ELIGIBILITY:
Inclusion Criteria:

* Males, Aged > 18 -< 55years old; weighing 55-75 kg
* Serum haemoglobin >10g/dl
* HIV negative status
* Written informed consent from the study subject.

Exclusion Criteria:

* Severe underlying conditions such as malnutrition (W/H <70%), clinically suspected cardiac, renal, or hepatic diseases, suspected AIDS, or severe injury.
* Presence of any concomitant illnesses such malaria, lower respiratory tract infections (LRTI), acute bloody or non-bloody diarrhoeas, or other as acute infections
* History of treatment with antimalarial drugs within the last 2 weeks
* History of treatment with aspirin or any non-steroidal-anti-inflammatory agent or trimethoprim and co-trimoxazole within the last 7 days.
* Any ongoing medication.
* Abnormal clinical chemistry or haematological finding
* Alcohol/drugs intake
* Any other reason in the recruiting clinician's opinion that makes the individual unsuitable for taking part in a clinical trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Clinical safety parameters:oral ulcers, GI tract disturbance,hematology, renal hepatic & other unsolicited safety AEs | 42 days

SECONDARY OUTCOMES:
Pharmacokinetics of Methotrexate assessed by repeated measurement of blood concentrations | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Nzila, Msc, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (1):
- Kenya Medical Research Institute, Center for Clinical Research, Nairobi, Nairobi County, Kenya

REFERENCES:
- [Result] Chilengi R, Juma R, Abdallah AM, Bashraheil M, Lodenyo H, Nyakundi P, Anabwani E, Salim A, Mwambingu G, Wenwa E, Jemutai J, Kipkeu C, Oyoo GO, Muchohi SN, Kokwaro G, Niehues T, Lang T, Nzila A. A phase I trial to evaluate the safety and pharmacokinetics of low-dose methotrexate as an anti-malarial drug in Kenyan adult healthy volunteers. Malar J. 2011 Mar 16;10:63. doi: 10.1186/1475-2875-10-63. PMID 21410944